CLINICAL TRIAL: NCT02802410
Title: Cross Sectional Study to Evaluate the Effects of Kinesio IQ-Tape, Kinesiotaping and no Taping on Muscle Activation and Reflex Activity During Climbing Stairs, Drop Jump and Running With 10, 12 and 15km/h
Brief Title: Cross Sectional Study to Evaluate Effects of Kinesiotaping on Muscle Activity During Climbing Stairs and Sport Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Heiner Baur (PhD), PD PhD, Bern University of Applied Sciences
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MSc - IQ-Tape
Record Dates: First submitted 2016-03-08; First posted 2016-06-16 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IQ-Tape (Experimental): IQ-application on leg muscles muscles
  Interventions: Device: IQ-Tape
- Kinesiotape (Experimental): Kinesiotape application on leg muscles
  Interventions: Device: Kinesiotape
- No-Tape (Experimental): No-Tape on leg muscles
  Interventions: Other: No-Tape

INTERVENTIONS:
Device: IQ-Tape — RMS-values of leg muscles at pre-activation (50ms) before ground-contact and post-activation 0-30ms and 30 - 150ms after ground-contact during drop-jump, running and stair climbing.
  Arms: IQ-Tape
Device: Kinesiotape — RMS-values of leg muscles at pre-activation (50ms) before ground-contact and post-activation 0-30ms and 30 - 150ms after ground-contact during drop-jump, running and stair climbing.
  Arms: Kinesiotape
Other: No-Tape — RMS-values of leg muscles at pre-activation (50ms) before ground-contact and post-activation 0-30ms and 30 - 150ms after ground-contact during drop-jump, running and stair climbing.
  Arms: No-Tape

SUMMARY:
This study aims to evaluate the effects of IQ-Tape, Kinesiotaping and no Taping on muscle activity during daily activity and sport activity.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* able to perform daily activities and sport performance

Exclusion Criteria:

* lower body and pelvic injuries
* fractures of the spine oder lower limb
* cardiac or neurological diseases

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Muscle activity of the quadriceps muscles during drop-jump, running and climbing stairs. | up to one week
  RMS-values of quadriceps muscles during, drop-jump, running with 10, 12 and 15km/h and stair climbing:
  pre-activation-phase: 50ms before ground-contact post-activation-phase: from 0 to 30ms and 30 to 150 ms after ground-contact

SECONDARY OUTCOMES:
Muscle activity of the hamstrings muscles during drop-jump, running and climbing stairs | up to one week
  RMS-values of hamstrings muscles during, drop-jump, running with 10, 12 and 15km/h and stair climbing:
  pre-activation-phase: 50ms before ground-contact post-activation-phase: from 0 to 30ms and 30 to 150 ms after ground-contact
Muscle activity of the soleus muscles during drop-jump, running and climbing stairs | up to me week
  RMS-values of soleus muscles during, drop-jump, running with 10, 12 and 15km/h and stair climbing:
  pre-activation-phase: 50ms before ground-contact post-activation-phase: from 0 to 30ms and 30 to 150 ms after ground-contact
Muscle activity of the tibialis muscles during drop-jump, running and climbing stairs | up to one week
  RMS-values of tibialis muscles during, drop-jump, running with 10, 12 and 15km/h and stair climbing:
  pre-activation-phase: 50ms before ground-contact post-activation-phase: from 0 to 30ms and 30 to 150 ms after ground-contact
Muscle activity of the gastrocnemius muscles during drop-jump, running and climbing stairs | up to one week
  RMS-values of gastrocnemius muscles during, drop-jump, running with 10, 12 and 15km/h and stair climbing:
  pre-activation-phase: 50ms before ground-contact post-activation-phase: from 0 to 30ms and 30 to 150 ms after ground-contact

CONTACTS AND LOCATIONS:
Locations (1):
- Bern University of Applied Sciences, Department Health, Bern, Switzerland